CLINICAL TRIAL: NCT04582188
Title: An Observational Study on the Prognostic Function of Early Coagulopathy in Sepsis Patients
Brief Title: The Early Coagulopathy for the Prognosis in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hua-Qing Shu, Associated Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: UHICU20201001
Record Dates: First submitted 2020-10-04; First posted 2020-10-09 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Sepsis; Coagulopathy; Outcome, Fatal
Keywords: Sepsis; Thrombomodulin; Thrombin-antithrombin complexe; Plasmin-α2-plasmin inhibitor complex; Tissue plasminogen activator-plasminogen activator inhibitor-1 complex; Mortality
MeSH Terms: conditions — Sepsis; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this cohort study, the parameters (TM, TAT, PIC, tPAIC, et al.) associated with the hemostatic system will be collected in sepsis patients when admitted to the Intensive Critical Unit. Parameters will be evaluated for their prognostic function of 28 days mortality.

DETAILED DESCRIPTION:
The object of this study is to find the early mortality prognostic biomarkers within the hemostatic system in sepsis patients. Blood samples will be collected from sepsis patients at admission. Parameters reflect endothelial injury, such as thrombomodulin (TM), tissue type plasminogen activator inhibitor complex (tPAIC), parameters reflect procoagulation condition, such as thrombin-antithrombin complex (TAT), and parameters reflect hyperfibrinolysis, such as plasmin-plasmin inhibitor complex (PIC) will be tested. Based on the results of these parameters, sepsis patients will be divided into coagulation parameter normal or abnormal groups. Twenty-eight days of mortality will be determined by patient follow-up. Regression analysis will be used to evaluate the relationship between these parameters and the mortality of sepsis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU of Union Hospital, Tongji Medical College, Huazhong University of Science and Technology from August 2020 to July 2022.
* Patients diagnosed with sepsis. The criteria for diagnosis is: 1. Infection or suspected infection; 2. SOFA score ≥ 2.
* Age interval: 18 years -- 80 years.
* Gender: unlimited.
* Signed informed consent form received.
* Results of the coagulation parameters tested within 24 hours after admission are available.

Exclusion Criteria:

* Pregnant and lactating women.
* With primary diseases that can cause thrombocytopenia or prolong prothrombin time, such as leukemia.
* Patients with severe liver dysfunction.
* Patients with anticoagulation or fibrinolysis medications within 72 hours before admission.
* Patients are in a procoagulation condition, such as VTE patients, protein C or protein S deficient individuals.
* Patients with chronic renal failure.
* Patients need ECMO therapy.
* Patients with severe cardiopulmonary diseases or nervous system diseases.
* Patients at the end-stage of disease.
* Patients without signed informed consent forms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients diagnosed with sepsis in the ICU of Union Hospital, Tongji Medical College, Huazhong University of Science and Technology.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-05 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
28-day all course mortality | 28 days from ICU-admission

SECONDARY OUTCOMES:
Length of stay | 28 days from ICU-admission
Length of using vasopressor | 28 days from ICU-admission